CLINICAL TRIAL: NCT00911235
Title: An Open-Label, Randomized, Two-Way Crossover Study To Evaluate The Effect Of Fluconazole, A Moderate CYP3A4 Inhibitor, On The Single-Dose Pharmacokinetics Of Fesoterodine In Healthy Subjects.
Brief Title: The Effect Of Fluconazole On Pharmacokinetics Of Fesoterodine In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A0221080
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Overactive Bladder With Symptoms of Frequency, Urgency, and Urge Urinary Incontinence
Keywords: The Effect Of Fluconazole On Pharmacokinetics Of Fesoterodine In Healthy Subjects
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — fesoterodine; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fesoterodine Alone (Experimental): Reference treatment
  Interventions: Drug: Fesoterodine
- fesoterodine plus fluconazole (Other): Test treatment
  Interventions: Drug: fesoterodine plus fluconazole

INTERVENTIONS:
Drug: Fesoterodine — Single 8 mg oral dose of fesoterodine
  Arms: Fesoterodine Alone
Drug: fesoterodine plus fluconazole — On Day 1, fluconazole (200 mg oral dose) will be given 1 hour before and approximately 11 hour following a single 8 mg oral dose of fesoterodine (fesoterodine SD). Fluconazole will also be administered 200 mg BID on the Day 2 (ie, at approximately 24 and 36 hours following the fesoterodine SD treatment given on Day 1)
  Arms: fesoterodine plus fluconazole

SUMMARY:
This study is designed to estimate the effect of fluconazole (200 mg BID for 2 days), a moderate CYP3A4 inhibitor on the pharmacokinetics of a single 8 mg oral dose of fesoterodine in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 18 and 55 years

Exclusion Criteria:

* Not healthy subjects. subjects with acute or chronic medical or psychiatric condition or laboratory abnormality

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
AUCinf and Cmax of 5-HMT | 3 days per period

SECONDARY OUTCOMES:
AUClast, Tmax and half-life of 5-HMT as data permit. | 3 days per period
Safety will be assessed by subjective symptoms/objective findings including physical examination findings, clinical safety laboratory assessments and adverse event monitoring. | 3 days per period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States